CLINICAL TRIAL: NCT01402050
Title: A Randomized Controlled Trial of Transcervical Foley Balloon Compared to Controlled Release Prostaglandin (Cervidil) for Labor Induction and Cervical Ripening in Term and Near Term Women
Brief Title: Foley Catheter Versus Cervidil for Induction of Labor at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-10-0012
Record Dates: First submitted 2011-04-08; First posted 2011-07-26 (Estimated); Results first posted 2020-02-06 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Labor Induction
Keywords: Time from the start of the induction to delivery
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLEY BALLOON (Active Comparator): Comparing foley balloon to cervidil for decreased time from the start of the induction process to delivery
  Interventions: Device: FOLEY BALLOON
- CERVIDIL (Active Comparator)
  Interventions: Drug: CERVIDIL (Dinoprostone)

INTERVENTIONS:
Drug: CERVIDIL (Dinoprostone) — INDUCTION OF LABOR
  Arms: CERVIDIL
Device: FOLEY BALLOON — INDUCTION OF LABOR
  Arms: FOLEY BALLOON

SUMMARY:
OBJECTIVE: To assess the efficacy of transcervical Foley catheter compared to controlled release prostaglandin (Cervidil™) for cervical ripening in term and near term women presenting for labor induction.

HYPOTHESIS: In term and near term women presenting for labor induction, transcervical Foley catheter will decrease the mean time from induction to delivery by six hours compared to controlled release prostaglandin (Cervidil™).

DETAILED DESCRIPTION:
BACKGROUND:

Induction of labor is performed in 25% of all women who present for delivery at the Banner Good Samaritan Medical Center (1). The commonality of labor induction is not only a local issue. The national cesarean rate has risen to 31.1%, which represents a 50% increase since 1996 (2). Part of the reason for this increase in the cesarean delivery rate is the pervasive use of labor induction. This risk can be mitigated with the use of cervical ripening agents when a cervix is unfavorable for induction. Both pharmacological (prostaglandin analogues) ripening agents and mechanical methods are utilized, but no single method has been shown to offer a significant advantage over the other methods. Many centers, including ours, have several different methods available, since each ripening method may have one or more unique contraindications for their use during labor induction.

One emerging modality for cervical ripening and labor induction has been transcervical Foley balloon catheter placement, which is thought to operate by mechanical dilation of the cervix. The modality has become popular in part due to its efficacy, safety and low cost. The most popular method of labor induction at Banner Good Samaritan Medical Center is a controlled release prostaglandin application (Cervidil™). This modality is expensive and may require more than one dose, thus increasing duration of labor induction and hospital costs. A thorough literature search was performed on PubMed with the search terms "foley" "labor induction" "prostaglandin E2 vaginal insert" from 1972 to 2009 and to date there have been no randomized trials comparing the efficacy of these two modalities for labor induction. Additionally, the clinical trials.gov site (www.clinicaltrials.gov) was searched and there are no active or previously complete studies of Cervidil™ compared to transcervical Foley balloon for labor induction. Therefore, we propose a randomized controlled clinical trial to evaluate the comparative efficacies of these two modalities for cervical ripening and labor induction in term and near term women.

METHODOLOGY:

All HIPAA and GCP regulations will be followed and IRB approval will be obtained.

This is a randomized controlled trial conducted at Banner Good Samaritan Medical Center (BGSMC) and Banner Desert Medical Center (BDMC) beginning February 1, 2010 and continuing until approximately 330 patients have been enrolled. Patients will be allocated by an online randomization system either to transcervical Foley catheter or controlled release prostaglandin (Cervidil™) in a 1:1 ratio. The Foley catheter used will be a 30cc/24 F. The Foley bulb is placed in the cervix and a balloon is filled with water to apply pressure to the cervix in order for the mechanical dilatation to occur. After the Foley catheter is placed, the RN will check (by gently tugging) the placement of the catheter every 2 hours until dislodged. Foley catheter will be removed either by spontaneous expulsion or after 12 hours if not expelled.

If the patient is randomized to the controlled release prostaglandin (Cervidil™) arm, a controlled release prostaglandin (Cervidil™) will be placed in the posterior fornix of the vagina to help ripen, or dilate and soften the cervix and removed after 12 hours. This medication may be repeated for an additional 12 hours per the physicians orders and standard of care procedures. The controlled release prostaglandin (Cervidil™) should be removed sooner if tachysystole (defined as more than 5 uterine contractions in 10 minutes) is noted.

After expulsion of the Foley catheter or after 12 hours in either group, oxytocin will be started according to the hospital's administration protocol. Otherwise, labor management will be at the discretion of the attending physician. Prophylactic antibiotics will not be administered unless indicated (GBS prophylaxis, chorioamnionitis develops during labor, etc).

A master subject list will be generated. Data collection forms will assign unique patient numbers starting with one and correlating with the master list. Data collection forms will not contain patient names, but the master list will have a number correlated with the patient ID. The data collection forms will collect demographic information including the date of birth for statistical analysis. All lists will be kept confidential and stored under locked conditions. The master list will be destroyed once the study is complete and the final report has been written.

Variables:

Outcomes:

1. Primary: Time from start of induction to delivery
2. Secondary:

   A. Proportion of patients delivered by 12 hours B. Proportion of patients delivered by 24 hours C. Proportion of patients delivered vaginally by 12 hours D. Proportion of patients delivered vaginally by 24 hours E. Chorioamnionitis (defined as a temperature of 38°C or higher and one of the following: maternal heart rate over 100, baseline fetal heart rate over 160, uterine tenderness, and/or purulent or foul-smelling cervical discharge) F. Endometritis (defined as a postpartum temperature of 38°C or higher on 2 or more occasions and no other source of fever) G. Overall cesarean rate H. Infection (Intrapartum, postpartum, cause of) I. Neonatal Information at delivery and discharge status (birth weight, apgars, cord pH, anomalies, NICU admission, other complications, neonatal death) J. Postpartum Information (Endometritis, Uterine tenderness, Maternal HR > 100 BMP, Purulent cervical discharge, wond complications, Ileus/Obstruction, Pneumonia, DVT/PTE (heparin treated) Intraperitoneal hematoma, Intraperitoneal abscess, UTI, Pyelonephritis, Maternal ICU admission, Maternal death) K. Date and time of Maternal and Neonatal discharge
3. Predictors:

A. Patient Demographics (date of birth, race, height, weight) B. Vital signs C. Maternal Comorbidities (Chronic Hypertension, Gestational Hypertension, Diabetes, Obesity or BMI) D. Induction Indications (Abnormal Antepartum Testing, Prior pregnancies, mode of deliveries, Pre-eclampsia, > 41 weeks gestation, Group Beta Strep status E. Physical Exam (Sterile vaginal exam, Membrane status) F. Study medication/device information (time of administration, removal, success of placement) G. Other induction medications (if indicated) H. Intrapartum antibiotics (if yes, reason for administration) I. Delivery data (date, time, mode of delivery)

STATISTICAL ANALYSIS: Descriptive statistics will be used, with continuous variables reported as means and standard deviations and categorical variables as percentages. T-tests will be used to analyze continuous variables and the Chi square test for categorical variables. Linear regression will be used to determine predictors of the primary outcome, and logistic regression for categorical outcomes. A two-tailed p < 0.05 will be considered significant.

SAMPLE SIZE CALCULATION: From review of the available literature evaluating these two modalites for labor induction (in separate studies), we make the following assumptions for our power calculation: 1. The mean time to delivery in the Cervidil group will be 24 hours. 2. The standard deviation for time to delivery in each group will be 15 hours. 3. A clinically significant decrease in the time to delivery in the Foley group is 6 hours (to a mean of 18 hours). With an alpha of 0.05 and 1-beta of 0.90, a sample size of 264 (132 in each group) is needed. Allowing a 20% cesarean delivery rate, so that a separate analysis can be performed for only those patients who delivered vaginally, the total number of women needed to be enrolled is 330.

INTERIM DATA ANALYSIS:

Because of the novel nature of this comparative induction regimen, an interim analysis and a futility analysis will be pursed when the first 100 of the study patients have been enrolled. The futility analysis will help direct trial progress.

A Data Safety Monitoring Board (DSMB) will be in place at the start of the study. The DSMB will comprise an independent obstetrician-gynecologist, a statistician and a bioethicist. It will regularly review SAE's.

It will also conduct an interim analysis when 100 subjects have had deliveries. Using the O'Brien-Fleming method, the p value for stopping the study due to superiority is 0.0051. At the final analysis, the remaining alpha for determining superiority is 0.0477. For the futility analysis, when 100 subjects have had a vaginal deliveries, a conditional power will be calculated. If the conditional power is < 0.20, then the study will be halted due to futility.

ELIGIBILITY:
Inclusion Criteria:

1. Cervix < 3 cm dilated. If 2cm dilated, must be < 80% effaced.
2. Gestational age ≥ 36 weeks by best obstetric estimate, and clinical management decision is delivery.
3. Singleton gestation
4. Cephalic presentation

Exclusion Criteria:

1. Regular uterine contractions (more frequent than every 5 minutes)
2. PROM
3. Prior transverse uterine incision or any obstetric contraindication to labor
4. Fever (defined as a temperature of 38°C or higher)
5. Lethal fetal anomalies (Labor induction is being performed, but there is no plan for fetal heart rate monitoring or cesarean delivery for fetal indications.)
6. Fetal death
7. Placenta previa
8. Suspected placental abruption or undiagnosed bleeding characterized as more than "spotting"
9. Non-reassuring fetal heart rate pattern
10. HIV

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 376 (Actual)
Dates: Start 2010-06; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique G Lin, MD, Principal Investigator — Obstetrix Medical Group
Locations (2):
- United States (2):
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Edwards RK, Szychowski JM, Berger JL, Petersen M, Ingersoll M, Bodea-Braescu AV, Lin MG. Foley catheter compared with the controlled-release dinoprostone insert: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1280-1287. doi: 10.1097/AOG.0000000000000238. PMID 24807327

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLEY BALLOON: Comparing Foley balloon to Cervidil for decreased time from the start of the induction process to delivery is the aim of this RCT.
  Subjects randomized into the Foley Balloon Arm received a Foley Balloon past the cervical os filled with 30 cc of sterile water, and catheter taped to inside of maternal thigh. Catheter was removed for any of the 5 reasons: expulsion, nonreasurring fetal heart rate tracing mandating placement of internal monitors, tachysystole, spontaneous membrane rupture, or 12 hours elapsed since placement.
  Key words: FOLEY BALLOON: INDUCTION OF LABOR
- CERVIDIL: CERVIDIL (Dinoprostone) Arm: Subjects randomized to this arm received dinoprostone controlled release vaginal insert (standard dosing Cervidil, 0.3mg/hour of dinoprostone over 12 hours). The vaginal insert was placed in the posterior fornix and was removed for any of the 5 reasons stated for the Foley catheter Arm description. Fetal heart rate and uterine contractions were continuously monitored per standard. Time of placement was noted as the time of Labor Induction initiation and time of delivery was noted as the end time of Labor Induction.
  Key word: INDUCTION OF LABOR
Period: Overall Study
Arm/Group | FOLEY BALLOON | CERVIDIL
Started | 185 | 191
Completed | 185 | 191
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLEY BALLOON | CERVIDIL | Total
Number analyzed (Participants) | 185 | 191 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (6.4) | 26.9 (5.9) | 27.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 191 | 376
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 81 | 168
  Black | 34 | 33 | 67
  Hispanic | 44 | 60 | 104
  Other | 20 | 17 | 37
Region of Enrollment [Number; unit: participants]
  United States | 185 | 191 | 376

OUTCOME MEASURES:

1. Primary Outcome: Time Of Start Of Induction Of Labor To Delivery
Description: The primary outcome variable was time (measured in hours) from first attempt at study agent placement to delivery. Time of placement of Labor Induction agent was noted as the time of Labor Induction initiation and time of delivery was noted as the end time of Labor Induction.
  There were no specific time points at which the outcomes were measured due to the uncertainty of the labor process. Total time duration of Labor induction was noted in hours.
  Key word: INDUCTION OF LABOR
Time Frame: Hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | FOLEY BALLOON | CERVIDIL
Number analyzed (Participants) | 185 | 191
hours | 21.6 [15.7 to 35.1] | 26.6 [19.0 to 37.8]

ADVERSE EVENTS:
Arm/Group | FOLEY BALLOON | CERVIDIL
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/191
Other Adverse Events (participants affected / at risk) | 0/185 | 2/191
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLEY BALLOON (N=185) | CERVIDIL (N=191)
Neonatal event (Gastrointestinal disorders) | 0 (0) | 2 (2) — Neonatal death due to pre-existing prenatally diagnosed diaphragmatic hernia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No